CLINICAL TRIAL: NCT05441813
Title: A Randomized, Open-label Study of Coconut Oil Mouth Rinse for Prophylaxis of Severe Oral Mucositis in Pediatric Patients Receiving Myeloablative Conditioning Regimens
Brief Title: Coconut Oil to Prevent Mouth Sores in Pediatric Patients Receiving High Dose Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCI-PED-BMT-MUC-001; Pro00061628 (Other: Advarra IRB); NCI-2024-06522 (Other: National Cancer Institute)
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis
Keywords: Prevention; Virgin Coconut Oil; Mouth Rinse
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care + virgin coconut oil (Experimental): Arm A: Standard of care + virgin coconut oil
  Interventions: Drug: Virgin Coconut Oil
- Standard of Care (No Intervention): Arm B: Standard of care

INTERVENTIONS:
Drug: Virgin Coconut Oil — Standard of care with the addition of virgin coconut oil mouth rinse
  Arms: Standard of care + virgin coconut oil

SUMMARY:
The purpose of this study is to learn if virgin coconut oil (VCO) mouth rinse can help prevent oral mucositis. The Study Investigator will compare standard of care mucositis prevention rinses with the VCO mouth rinse added to the standard of care mucositis prevention rinses. The severity of oral mucositis between the 2 groups will be evaluated. Some of the standard of care rinses that can be used to prevent mucositis are normal saline, Benadryl (diphenhydramine), Mylanta, lidocaine, or other combinations.

DETAILED DESCRIPTION:
This is a randomized, open-label study. The target population is patients ≥ 7 years to 26 years at time of consent who are planning to undergo myeloablative conditioning regimens in preparation HSCT. The study will be conducted at Levine Children's Hospital, Levine Children's Cancer and Blood Disorders Clinic and Atrium Health. Subjects will be screened and consented within 28 days prior to admission. The planned treatment period for Arm A (standard of care with the addition of VCO mouth rinses) or Arm B (standard of care) will begin at the start of subject's admission for conditioning, followed by transplant event with day of transplant defined as Day 0 and continue through Day +45 following transplant or hospital discharge, whichever comes first. A Safety Follow Up Visit will occur no sooner than 30 days from last study drug treatment

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all the following applicable inclusion criteria to participate in this study:

1. Written informed consent, HIPAA authorization for release of personal health information, and assent, when applicable from the subject, parent, or legal guardian.
2. Age greater than or equal to 7 years to 26 years at the time of consent
3. Patients planning to undergo myeloablative conditioning regimens in preparation for HSCT
4. ECOG Performance Status of less than or equal to 2 or Lansky/Karnofsky Performance Status of greater than or equal to 50 within 7 days prior to date of enrollment.
5. No evidence of mouth lesions at time of enrollment
6. Ability of the subject and parent/caregiver to understand and comply with study procedures for the entire length of the study
7. Able and willing to swish/spit the oral formulation

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

1. Allergy to tree nuts
2. Planned discharge home prior to engraftment
3. Using coconut oil mouth rinses within 30 days prior to enrollment
4. Using additional mouthcare regimens, other than those allowed in the institutional SOP, prior to admission with a plan to continue use during admission
5. Patient has undergone HSCT within the last 90 days prior to admission

Ages: 7 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2036-07 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Severity of Mucositis | Day 45
  Using Area Under the Curve (AUC) of the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 mucositis oral grading scale. This is a 5-point ordered-categorical scale ranging from 1 (asymptomatic or mild symptoms) to 5 (death). For subjects not experiencing oral mucositis, a severity grade of zero will be assigned.

SECONDARY OUTCOMES:
Average Daily Caloric Intake | Day 45
  Oral intake will be calculated quantitatively for each subject during the on-treatment period.
Total Parenteral Nutrition (TPN) | Day 45
  TPN or hyperalimentation will be calculated quantitatively for each subject as the proportion of days during the on-treatment period that aggressive nutrition support was utilized.
Opioid Use | Day 45
  Daily opioid use will be calculated quantitatively for each subject in terms of their average Morphine Equivalent Daily Dose (MEDD)
Time to CTCAE Mucositis Grade > 2 | Day 45
  The duration of time (in days) from the initiation of study treatment until the day of the first occurrence of a CTCAE mucositis grade exceeding 2. The CTCAE mucositis grade is a 5-point ordered-categorical scale ranging from 1 (asymptomatic or mild symptoms) to 5 (death). For subjects who do not report a grade exceeding 2, time to CTCAE mucositis grade >2 will be censored at the date of the last completed CTCAE evaluation.
Daily Incidence of Optional Mouth Rinses | Day 45
  Proportion of days during the on-treatment period that optional oral rinse was used.
Incidence and type of oral viral infections | Day 45
  Incidence and type of oral viral infections
Length of Hospitalization | Day 45
  Length of stay will be calculated for each subject as the number of days from admission date to discharge date +1.
Days to Absolute Neutrophil Count (ANC) Engraftment | Day 45
  Days to engraftment will be calculated for each subject as the number of days from Hematopoietic Stem Cell Transplantation (HSCT) to ANC recovery per Center for International Blood and Marrow Transplantation Research (CIBMTR) definition

OTHER OUTCOMES:
Oral Rinse Utilization | Day 45
  Reported as a percent of utilization

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Huddle, MSN, RDN, CSPCC, LDN, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Levine Children's Hospital, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No